CLINICAL TRIAL: NCT06340256
Title: Comparative Study Between Continuous Spinal Anesthesia Versus Epidural Anesthesia in Geriatric Patients Undergoing Major Hip Surgery
Brief Title: Continuous Spinal Anesthesia Versus Epidural Anesthesia in Geriatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Professor Of Anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB0000871253
Record Dates: First submitted 2024-03-23; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Epidural Catheter

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ! (Active Comparator): Continuous spinal anesthesia
  Interventions: Other: Continuous spinal anesthesia
- Group 2 (Active Comparator): Continuous epidural anesthesia
  Interventions: Other: Continuous epidural anesthesia

INTERVENTIONS:
Other: Continuous spinal anesthesia — The Catheter will be then fed over the needle into the intrathecal space and Inserted 3cm cephalad into the subarachnoid space.The spinal needle and the modified Tuohy needle will be then removed, and a Luer connector and A filter previously filled with the anesthetic solution will be attached to the Catheter (priming volume 0.6ml). Plain bupivacaine 0.5% in 20ml vials will Be used CSA group received 1 ml(5 mg) of plain bupivacaine (0.5%) Together with fentanyl l25μg injected via the catheter at a rate of 0.2ml/15s. The level of the resulting sensory blockade will be tested using pin prick.
  Arms: Group !
Other: Continuous epidural anesthesia — The needle is advanced until the epidural space is identified by the loss-of-resistance technique, and then a 20G catheter is inserted 3 cm cephalad into the epidural space. a test dose of 3ml of 2% lignocaine with adrenaline (1:200000) will be injected into the catheter. Three minutes later, 10 ml of plain bupivacaine (0.5%) together with fentanyl l50μg will be injected via the catheter.
  Arms: Group 2

SUMMARY:
60 patients aged older than 60 years, American Society of Anesthesiologists (ASA) class II or III and scheduled for major hip surgery will be randomized, in to two groups anesthetized using continuous spinal anesthesia or using continuous epidural anesthesia.

DETAILED DESCRIPTION:
60 patients aged older than 60 years, American Society of Anesthesiologists (ASA) class II or III and scheduled for major hip surgery will be randomized, in to two groups anesthetized using continuous spinal anesthesia or using continuous epidural anesthesia.

In continuous spinal anesthesia group 22 G catheter with priming volume0.1m The Catheter will be then fed over the needle into the intrathecal space and Inserted 3cm cephalad into the subarachnoid space.The spinal needle and the modified Tuohy needle will be then removed, and a Luer connector and A filter previously filled with the anesthetic solution will be attached to the Catheter (priming volume 0.6ml). Plain bupivacaine 0.5% in 20ml vials will Be used CSA group received 1 ml(5 mg) of plain bupivacaine (0.5%) Together with fentanyl l25μg injected via the catheter at a rate of 0.2ml/15s. The level of the resulting sensory blockade will be tested using pin prick.

Continuous epidural anesthesia Group A Perifix 401filter epidural set.It is composed of Tuohy epidural needle1.3×80 mm (18G);an epidural catheter with three lateral openings 0.85×0.45×1000 mm (20G); loss-of-resistance syringe, 10 ml; a Perifix flat filter 0.2μm; and Perifix screw connector. The needle is advanced until the epidural space is identified by the loss-of-resistance technique, and then a 20G catheter is inserted 3 cm cephalad into the epidural spac e. a test dose of 3ml of 2% lignocaine with adrenaline (1:200000) will be injected into the catheter. Three minutes later, 10 ml of plain bupivacaine (0.5%) together with fentanyl l50μg will be injected via the catheter. If the sensory blockade don't reach T10 within 20 min of the administration of the initial dose, additional doses of 5 ml of plain bupivacaine 0.5% will be injected epidurally every10 min until the level of T10 or amaximum of 25 ml of plain bupivacaine 0.5 % will be achieved. If the sensory blockade don't not reach T10, anesthetic failure will be considered, and the patients will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* patients aged older than 60 years
* American Society of Anesthesiologists (ASA) class II or III
* scheduled for major hip surgery

Exclusion Criteria:

* -Refusal
* Infection at the injection site
* Spinal deformity
* Neuropathy
* Allergy to local anesthetics
* Coagulopathy

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Hemodynamic changes | during the surgery
  mean arterial blood pressure

SECONDARY OUTCOMES:
Patient satisfaction | immediately after the surgery
  At the end of the surgery by verbal rating score

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Thabet, Principal Investigator — Al-Azhar Faculty of Medicine
Locations (1):
- Al-Azhar Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Imbelloni LE, Gouveia MA, Cordeiro JA. Continuous spinal anesthesia versus combined spinal epidural block for major orthopedic surgery: prospective randomized study. Sao Paulo Med J. 2009 Jan;127(1):7-11. doi: 10.1590/s1516-31802009000100003. PMID 19466288